CLINICAL TRIAL: NCT00670111
Title: Restoration of Chronotropic Competence in Heart Failure Patients With Normal Ejection Fraction
Acronym: RESET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrollment
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RESET
Record Dates: First submitted 2008-04-23; First posted 2008-05-01 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure
Keywords: Heart failure; exercise capacity; ejection fraction; Heart failure normal ejection fraction
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAP On then Off at 1 month visit (Experimental): 1. Rate Adaptive Pacing (RAP) On for first cardiopulmonary exercise test (CPX) at one month.
  2. Rate Adaptive Pacing (RAP) Off for second cardiopulmonary exercise test (CPX) at one month.
  Interventions: Device: Insignia Plus / Ultra (Guidant/Boston Scientific)
- RAP Off then On at 1 month visit (Experimental): 1. Rate Adaptive Pacing (RAP) Off for first cardiopulmonary exercise test (CPX) at one month.
  2. Rate Adaptive Pacing (RAP) On for second cardiopulmonary exercise test (CPX) at one month.
  Interventions: Device: Insignia Plus / Ultra (Guidant/Boston Scientific)

INTERVENTIONS:
Device: Insignia Plus / Ultra (Guidant/Boston Scientific) — Cardiac pacing using any Guidant/Boston Scientific Implantable Pacemaker System with rate-modulation and any compatible intracardiac lead system.
  Other Names: Guidant or Boston Scientific implantable pacemakers

SUMMARY:
This study will look at how pacing your heart may assist your daily activities and how you are feeling.

DETAILED DESCRIPTION:
RESET is a multicenter trial that will assess the effect of pacing in heart failure patients with a normal ejection fraction (or diastolic heart failure). The purpose of the RESET study is to evaluate the effect of pacing on exercise capacity and quality of life in this heart failure population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are in sinus rhythm
* Patients who are on stable medical therapy
* Patients who exhibit signs and symptoms of heart failure, New York Heart Association (NYHA) Class II or III
* Patients who have experienced a hospitalization for decompensated heart failure; treatment for pulmonary congestion or volume overload; chronic treatment with a loop diuretic; or a brain natriuretic peptide (BNP) > 125 ng/l.
* Left ventricular ejection fraction (LVEF) ≥ 50%

Exclusion Criteria:

* Patients with persistent atrial fibrillation or atrial flutter
* Patients who are in complete heart block
* Patients who have experienced a recent myocardial infarction (MI) or have unstable angina or require cardiac surgery or other procedures
* Patients who have severe heart valve disease or valve replacement
* Patients with a contraindication for a pacemaker system
* Patients who have a neuromuscular, orthopedic or other non-cardiac condition that prevents patient from exercise testing
* Patients who have infiltrative or hypertrophic cardiomyopathy
* Patients who have known severe pulmonary disease
* Patients with uncontrolled diabetes or blood pressure (systolic blood pressure (SBP) > 160 mmHg or diastolic blood pressure (DBP) > 95 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Kass, M.D., Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - Cardiovascular Associates of Northeast Arkansas, Jonesboro, Arkansas
  - Cardiovascular Associates, Louisville, Kentucky
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Mayo Clinic Foundation, Rochester, Minnesota
  - Tyler CV Consultants - Trinity Mother Frances, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kass DA, Kitzman DW, Alvarez GE. The restoration of chronotropic competence in heart failure patients with normal ejection fraction (RESET) study: rationale and design. J Card Fail. 2010 Jan;16(1):17-24. doi: 10.1016/j.cardfail.2009.08.008. Epub 2009 Oct 7. PMID 20123314

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment, patients were had an exercise test to determine chronotropic incompetence (CI). If patients were not CI, they were deemed a Testing Failure and withdrawn from the study. CI patients that were then implanted with a pacemaker were randomized to the order of their Rate Adaptive Pacing therapy for the 2 one month exercise tests.
Groups:
- Rate Adaptive Pacing (RAP) On Then Off: Rate Adaptive Pacing (RAP) On for first cardiopulmonary exercise test (CPX) at one month, then RAP-Off for second CPX at one month.
- Rate Adaptive Pacing (RAP) Off Then On: Rate Adaptive Pacing (RAP) Off for first cardiopulmonary exercise test (CPX) at one month, then RAP-On for second CPX at one month.
- Non-Randomized Patients: Only implanted patients were randomized. All other patients fall into this group.
Period: Enrollment to One Month
Arm/Group | Rate Adaptive Pacing (RAP) On Then Off | Rate Adaptive Pacing (RAP) Off Then On | Non-Randomized Patients
Started | 5 | 8 | 19
Completed | 4 | 8 | 0
Not Completed | 1 | 0 | 19
Not completed — Testing Failure | 0 | 0 | 13
Not completed — Ebrolled Patients but not Implanted | 0 | 0 | 6
Not completed — Physician Decision | 1 | 0 | 0
Period: One Month Period A
Arm/Group | Rate Adaptive Pacing (RAP) On Then Off | Rate Adaptive Pacing (RAP) Off Then On | Non-Randomized Patients
Started | 4 | 8 | 0
Completed | 4 | 8 | 0
Not Completed | 0 | 0 | 0
Period: One Month Period B
Arm/Group | Rate Adaptive Pacing (RAP) On Then Off | Rate Adaptive Pacing (RAP) Off Then On | Non-Randomized Patients
Started | 4 | 8 | 0
Completed | 4 (4 patients in this group completed the 1 month visit; 0 had data eligible for endpoint analysis.) | 8 (8 patients in this group completed the 1 month visit; 6 had data eligible for endpoint analysis.) | 0
Not Completed | 0 | 0 | 0
Period: One Month to Six Months
Arm/Group | Rate Adaptive Pacing (RAP) On Then Off | Rate Adaptive Pacing (RAP) Off Then On | Non-Randomized Patients
Started | 4 | 8 | 0
Completed | 4 (4 patients in this group completed the 1 month visit; 0 had data eligible for endpoint analysis.) | 8 (8 patients in this group completed the 1 month visit; 4 had data eligible for endpoint analysis.) | 0
Not Completed | 0 | 0 | 0
Period: Six Months to Twelve Months
Arm/Group | Rate Adaptive Pacing (RAP) On Then Off | Rate Adaptive Pacing (RAP) Off Then On | Non-Randomized Patients
Started | 4 | 8 | 0
Completed | 4 | 8 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants were "RAP On" for months 1 through 6. All participants were 'Rap On' for months 6 to 12.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rate Adaptive Pacing (RAP) On Then Off | Rate Adaptive Pacing (RAP) Off Then On | Non-Randomized Patients | Total
Number analyzed (Participants) | 5 | 8 | 19 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 5 | 8
  >=65 years | 4 | 6 | 14 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (7.1) | 65.8 (12.1) | 68.1 (11.0) | 67.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 10 | 18
  Male | 2 | 3 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 19 | 32

OUTCOME MEASURES:

1. Primary Outcome: Peak Volume of Oxygen Uptake (Peak VO2) - Rate Adaptive Pacing (RAP) On at One Month vs. Rate Adaptive Pacing (RAP) Off at One Month.
Description: Randomized therapy order cross-over comparison at 1 month post-implant. Each patient evaluated for endpoint with and without RAP therapy at this time.
Time Frame: 1 month post implant
Population: The following were required for a patient's dataset to be included in the analysis:
  1. 2 CPX tests had to be performed at 1M (RAP On & RAP Off),
  2. Each 1M CPX test had to result in RER ≥ 1.05,
  3. Trending data from the disk had to have been obtained during each 1M CPX test.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Rate Adaptive Pacing (RAP) On at One Month: Rate Adaptive Pacing (RAP) On for cardiopulmonary exercise test (CPX) at one month.
- Rate Adaptive Pacing (RAP) Off at One Month: Rate Adaptive Pacing (RAP) Off for cardiopulmonary exercise test (CPX) at one month.
Arm/Group | Rate Adaptive Pacing (RAP) On at One Month | Rate Adaptive Pacing (RAP) Off at One Month
Number analyzed (Participants) | 6 | 6
ml/kg/min | 12.47 (2.02) | 12.79 (2.14)

2. Secondary Outcome: Peak Volume of Oxygen Uptake (Peak VO2) - Rate Adaptive Pacing (RAP) On at Six Months vs. Rate Adaptive Pacing (RAP) Off at One Month.
Description: Each patient had RAP therapy On from one through six months. This endpoint evaluated Peak VO2 measured at 6 months (RAP On) vs. Peak VO2 measured at 1 month without RAP therapy (RAP Off).All participants were "RAP On" for months 1 through 6. All participants were 'Rap On' for months 6 to 12.
Time Frame: 6 months post implant
Population: The following were required for a patient's dataset to be included in the analysis:
  1. 2 CPX tests had to be performed (1M with RAP Off, 6M with RAP On [RAP was On from 1M to 6M]),
  2. Each CPX test had to result in RER ≥ 1.05,
  3. Trending data from the disk had to have been obtained during each CPX test.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Rate Adaptive Pacing (RAP) On at Six Months: Rate Adaptive Pacing (RAP) On for first cardiopulmonary exercise test (CPX) at one month, then RAP-Off for second CPX at one month.
- Rate Adaptive Pacing (RAP) Off at One Month: Rate Adaptive Pacing (RAP) Off for first cardiopulmonary exercise test (CPX) at one month, then RAP-On for second CPX at one month.
Arm/Group | Rate Adaptive Pacing (RAP) On at Six Months | Rate Adaptive Pacing (RAP) Off at One Month
Number analyzed (Participants) | 4 | 4
ml/kg/min | 12.04 (1.74) | 13.09 (2.35)

ADVERSE EVENTS:
Time Frame: Entire study (twelve months)
Description: Adverse events were collected for all enrolled patients.
Groups:
- All Implanted Patients: All patients from the RAP On then Off group and from the RAP Off then On group.
- Non-Randomized Patients: Only implanted patients were randomized. All other patients fall into this group. Adverse events were collected for all subjects, also for non-randomized patients.
Arm/Group | All Implanted Patients | Non-Randomized Patients
Serious Adverse Events (participants affected / at risk) | 7/13 | 0/19
Other Adverse Events (participants affected / at risk) | 10/13 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Implanted Patients (N=13) | Non-Randomized Patients (N=19)
Cerebrovascular accident (CVA) (Vascular disorders) | 1 (1) | 0 (0)
Chronic cervical spondylosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Genitourinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 4 (7) | 0 (0)
Hematological - Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0)
Integumentary (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Knee replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lead Dislodgment, Right Atrial (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia, lingular (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rate response inappropriate - Pulse generator (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Implanted Patients (N=13) | Non-Randomized Patients (N=19)
Adverse reaction - Rash from ECG leads (Surgical and medical procedures) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0)
Chest pain (Cardiac disorders) | 3 (3) | 0 (0)
Chest pain - due to acid reflux (Cardiac disorders) | 1 (1) | 0 (0)
Coughing, Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 2 (4) | 0 (0)
Integumentary - Herpes zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Integumentary - Skin reaction to adhesive (Surgical and medical procedures) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Oversensing, Right Atrial (Cardiac disorders) | 1 (1) | 0 (0)
Rapid heart rate (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early study termination leading to small numbers of subjects analyzed and an inability to test study hypothesis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other